CLINICAL TRIAL: NCT04568148
Title: COVID-19 Biorepository
Status: Active, not recruiting | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Leslie Spikes, MD, Assistant Professor, University of Kansas Medical Center
Other Study IDs: STUDY#00145602
Record Dates: First submitted 2020-04-15; First posted 2020-09-29 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Covid-19; SARS-CoV 2; Coronavirus; COVID
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Biospecimens to be collected include serum and plasma. Blood samples will be collected, processed, aliquoted, and stored at -80°C. A portion of the blood samples will be kept for DNA and RNA isolation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Establish a COVID-19 biorepository to aid in developing our knowledge of the disease.

DETAILED DESCRIPTION:
While SARS-CoV-2 has some similarities to the SARS-CoV pathogen that led to an epidemic in 2002 and 2003, there is much about the epidemiology, pathogenesis, clinical presentation, diagnosis, and treatment of the novel virus that remains unknown.3 Additional research is needed to explore the nature of the virus, its spectrum of disease, and potential therapies to combat its spread. The aim of this project will be to establish a biorepository of blood samples from patients infected with SARS-CoV-2 that can then be used by investigators to expand our understanding of COVID-19 and its treatment and, in turn, improve patient outcomes.

The COVID-19 biorepository will accomplish the following specific aims:

1. Establish a collection of biospecimens from patients with COVID-19.
2. Establish a link between biospecimens and longitudinal individual patient data, which will be collected and stored in RedCap.
3. Provide biospecimens and unique patient data to researchers investigating COVID-19. Separate IRB approval will be needed for these studies.

ELIGIBILITY:
Inclusion Criteria:

* The participant is a patient at TUKHS or has agreed to participate in a study approved by the KUMC Human Research Protection Program (HRPP).
* The participant has a diagnosis of COVID-19 confirmed by COVID-19 PCR.
* Patient is 18 years of age or older.

Exclusion Criteria:

* Participant declines to participate (living patients only)
* Participant or healthcare surrogate is unable to provide informed consent (living patients only)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: COVID-19-positive patients
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Biospecimen Collection | From Enrollment to 3 Months
  Establish a collection of biospecimens from patients with COVID-19.
Establishing Connections | From Enrollment to 3 Months
  Establish a link between biospecimens and longitudinal individual patient data
Continuing COVID Research | From Enrollment to 3 Months
  Provide biospecimens and unique patient data to researchers investigating COVID-19

CONTACTS AND LOCATIONS:
Overall Officials: Leslie A Spikes, MD, Principal Investigator — Assistant Professor of Medicine
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided